CLINICAL TRIAL: NCT04996797
Title: A Phase 2, Multi-Center, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Induction Therapy With PRA023 in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Phase 2 Safety and Efficacy Study of Tulisokibart (MK-7240/PRA023) in Subjects With Moderately to Severely Active Ulcerative Colitis (MK-7240-005)
Acronym: ARTEMIS-UC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prometheus Biosciences, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR200-102; MK-7240-005 (Other: MSD ID); PRA023 (Other: Prometheus Biosciences); 2023-509741-12-00 (Registry Identifier: EU CT); U1111-1309-6078 (Registry Identifier: UTN); 2021-000091-11 (EudraCT Number)
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis
Keywords: ARTEMIS-UC; ARTEMIS; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative; Severe combined immunodeficiency with sensitivity to ionizing radiation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Cohort 1 Tulisokibart (Experimental): Participants who are CDx+ and CDx- will receive tulisokibart administered by intravenous (IV) infusion at 1000 mg on Day 1, Week 0, and 500 mg on the first day of Weeks 2, 6, and 10. After the completion of the 12-week induction, all participants have the option to continue in the open-label extension for up to 170 weeks.
  Interventions: Drug: Tulisokibart
- Cohort 1 Placebo (Placebo Comparator): Participants who are CDx+ and CDx- will receive placebo administered by intravenous (IV) infusion on Day 1, Week 0 and the first day of Weeks 2, 6, and 10. After the completion of the 12-week induction, all participants have the option to continue in the open-label extension for up to 170 weeks.
  Interventions: Other: Placebo
- Cohort 2 Tulisokibart (Experimental): Participants who are CDx+ will receive tulisokibart administered by intravenous (IV) infusion at 1000 mg on Day 1, Week 0 and 500 mg on the first day of Weeks 2, 6, and 10. After the completion of the 12-week induction, all participants have the option to continue in the open-label extension for up to 170 weeks.
  Interventions: Drug: Tulisokibart; Device: Companion Diagnostic (CDx) Testing
- Cohort 2 Placebo (Placebo Comparator): Participants who are CDx+ will receive placebo administered by intravenous (IV) infusion on Day 1, Week 0 and the first day of Weeks 2, 6, and 10. After the completion of the 12-week induction, all participants have the option to continue in the open-label extension for up to 170 weeks.
  Interventions: Device: Companion Diagnostic (CDx) Testing; Other: Placebo

INTERVENTIONS:
Drug: Tulisokibart — Administered by IV infusion
  Other Names: MK-7240; PRA023
  Arms: Cohort 1 Tulisokibart; Cohort 2 Tulisokibart
Device: Companion Diagnostic (CDx) Testing — PRA023 CDx Genotyping Assay
  Arms: Cohort 2 Placebo; Cohort 2 Tulisokibart
Other: Placebo — Placebo administered by IV infusion
  Arms: Cohort 1 Placebo; Cohort 2 Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of tulisokibart in participants with moderately to severely active Ulcerative Colitis (UC). After the completion of the 12-week induction, all participants have the option to continue in the open-label extension for up to 170 weeks.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Confirmed diagnosis of ulcerative colitis (UC)
* Has moderately to severely active UC as defined by 3-component Modified Mayo score
* Must have corticosteroid dependence or have had no response, insufficient response, loss of response, and/or intolerance to at least one of the following therapies: corticosteroid, immunosuppressants, or an approved anti-tumor necrosis factor (anti-TNF), anti-integrin, anti-interleukin 12/23 (anti-IL12/23), Janus kinase (JAK) inhibitor, Sphingosine 1-phosphate receptor (S1PR) modulator.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has diagnosis of Crohn's disease or indeterminate colitis
* Has current evidence of fulminant colitis, toxic megacolon, bowel perforation, total proctocoloectomy or partial colectomy
* Has current or impending need for colostomy or ileostomy
* Has had surgical bowel resection within 3 months before screening
* Has past or current evidence of definite low-grade or high-grade colonic dysplasia not completely removed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2025-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (82):
- United States (27):
  - Prometheus Biosciences Selected Center, Mobile, Alabama
  - Prometheus Biosciences Selected Site, Phoenix, Arizona
  - Prometheus Biosciences Selected Site, Sun City, Arizona
  - Prometheus Biosciences Selected Site, Los Angeles, California
  - Prometheus Biosciences Selected Site, San Diego, California
  - Prometheus Biosciences Selected Site, Bristol, Connecticut
  - Prometheus Biosciences Selected Site, Atlanta, Georgia
  - Prometheus Biosciences Selected Site, Arlington Heights, Illinois
  - Prometheus Biosciences Selected Site, Glenview, Illinois
  - Prometheus Biosciences Selected Site, Gurnee, Illinois
  - Prometheus Biosciences Selected Site, Kansas City, Kansas
  - Prometheus Biosciences Selected Site, Liberty, Kansas
  - Prometheus Biosciences Selected Site, Baton Rouge, Louisiana
  - Prometheus Biosciences Selected Site, Chevy Chase, Maryland
  - Prometheus Biosciences Selected Site, Chesterfield, Michigan
  - Prometheus Biosciences Selected Site, Lebanon, New Hampshire
  - Prometheus Biosciences Selected Site, New York, New York
  - Prometheus Biosciences Selected Site, Dublin, Ohio
  - Prometheus Biosciences Selected Site, Germantown, Tennessee
  - Prometheus Biosciences Selected Site, Bedford, Texas
  - Prometheus Biosciences Selected Site, Lubbock, Texas
  - Prometheus Biosciences Selected Site, Mansfield, Texas
  - Prometheus Biosciences Selected Site, San Antonio, Texas
  - Prometheus Biosciences Selected Site, Southlake, Texas
  - Prometheus Biosciences Selected Site, Tyler, Texas
  - Prometheus Biosciences Selected Site, Charlottesville, Virginia
  - Prometheus Biosciences Selected Site, Tacoma, Washington
- Australia (8):
  - Prometheus Biosciences Selected Site, Woodville, Adelaide
  - Prometheus Biosciences Selected Site, Kingswood, New South Wales
  - Prometheus Biosciences Selected Site, Old Toongabbie, New South Wales
  - Prometheus Biosciences Selected Site, South Brisbane, Queensland
  - Prometheus Biosciences Selected Site, Woolloongabba, Queensland
  - Prometheus Biosciences Selected Site, Adelaide, South Australia
  - Prometheus Biosciences Selected Site, Fitzroy, Victoria
  - Prometheus Biosciences Selected Site, Melbourne, Victoria
- Belgium (2):
  - Prometheus Biosciences Selected Site, Leuven
  - Prometheus Biosciences Selected Site, Liège
- Canada (4):
  - Prometheus Biosciences Selected Site, Calgary, Alberta
  - Prometheus Biosciences Selected Site, Vancouver, British Columbia
  - Prometheus Biosciences Selected Site, Halifax, Nova Scotia
  - Prometheus Biosciences Selected Site, North York, Ontario
- Czechia (4):
  - Prometheus Biosciences Selected Site, Brno
  - Prometheus Biosciences Selected Site, Hradec Králové
  - Prometheus Biosciences Selected Site, Olomouc
  - Prometheus Biosciences Selected Site, Slaný
- France (6):
  - Prometheus Biosciences Selected Site, Clichy
  - Prometheus Biosciences Selected Site, Lille
  - Prometheus Biosciences Selected Site, Nice
  - Prometheus Biosciences Selected Site, Pierre-Bénite
  - Prometheus Biosciences Selected Site, Saint-Priest-en-Jarez
  - Prometheus Biosciences Selected Site, Vandœuvre-lès-Nancy
- Prometheus Biosciences Selected Site, Tbilisi, Georgia
- Hungary (4):
  - Prometheus Biosciences Selected Site, Győr, Győr-Moson-Sopron
  - Prometheus Biosciences Selected Site, Békéscsaba
  - Prometheus Biosciences Selected Site, Budapest
  - Prometheus Biosciences Selected Center, Budapest
- Israel (5):
  - Prometheus Biosciences Selected Site, Afula
  - Prometheus Biosciences Selected Site, Beersheba
  - Prometheus Biosciences Selected Site, Holon
  - Prometheus Biosciences Selected Site, Jerusalem
  - Prometheus Biosciences Selected Site, Petah Tikva
- Italy (3):
  - Prometheus Biosciences Selected Site, Bologna, Emilia-Romagna
  - Prometheus Biosciences Selected Site, Milan, Milan
  - Prometheus Biosciences Selected Site, Roma, Rome
- Poland (16):
  - Prometheus Biosciences Selected Site, Poznan, Greater Poland Voivodeship
  - Prometheus Biosciences Selected Site, Włocławek, Kuuavian-Pomeranian
  - Prometheus Biosciences Selected Site, Krakow, Lesser Poland Voivodeship
  - Prometheus Biosciences Selected Site, Wroclaw, Lower Silesian Voivodeship
  - Prometheus Biosciences Selected Site, Warsaw, Masovia
  - Prometheus Biosciences Selected Site, Katowice, Silesian
  - Prometheus Biosciences Selected Site, Krakow
  - Prometheus Biosciences Selected Site, Lodz
  - Prometheus Biosciences Selected Site, Lublin
  - Prometheus Biosciences Selected Site, Rzeszów
  - Prometheus Biosciences Selected Site, Sopot
  - Prometheus Biosciences Selected Site, Szczecin
  - Prometheus Biosciences Selected Site, Torun
  - Prometheus Biosciences Selected Site #2, Warsaw
  - Prometheus Biosciences Selected Site, Warsaw
  - Prometheus Biosciences Selected Site, Wroclaw
- United Kingdom (2):
  - Prometheus Biosciences Selected Site, Prescot, Merseyside
  - Prometheus Biosciences Selected Sites, London

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Sands BE, Feagan BG, Peyrin-Biroulet L, Danese S, Rubin DT, Laurent O, Luo A, Nguyen DD, Lu J, Yen M, Leszczyszyn J, Kempinski R, McGovern DPB, Ma C, Ritter TE, Targan S; ARTEMIS-UC Study Group. Phase 2 Trial of Anti-TL1A Monoclonal Antibody Tulisokibart for Ulcerative Colitis. N Engl J Med. 2024 Sep 26;391(12):1119-1129. doi: 10.1056/NEJMoa2314076. PMID 39321363
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26158&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with moderately to severely active ulcerative colitis were enrolled.
Groups:
- Cohort 1 Tulisokibart: Participants who were CDx+ and CDx- received tulisokibart administered by intravenous (IV) infusion at 1000 mg on Day 1, Week 0, and 500 mg on the first day of Weeks 2, 6, and 10. After the completion of the 12-week induction, all participants have the option to continue in the open-label extension for up to 170 weeks.
- Cohort 1 Placebo: Participants who were CDx+ and CDx- received placebo administered by intravenous (IV) infusion on Day 1, Week 0 and the first day of Weeks 2, 6, and 10. After the completion of the 12-week induction, all participants have the option to continue in the open-label extension for up to 170 weeks.
- Cohort 2 Tulisokibart: Participants who were CDx+ received tulisokibart administered by intravenous (IV) infusion at 1000 mg on Day 1, Week 0 and 500 mg on the first day of Weeks 2, 6, and 10. After the completion of the 12-week induction, all participants have the option to continue in the open-label extension for up to 170 weeks.
- Cohort 2 Placebo: Participants who were CDx+ received placebo administered by intravenous (IV) infusion on Day 1, Week 0 and the first day of Weeks 2, 6, and 10. After the completion of the 12-week induction, all participants have the option to continue in the open-label extension for up to 170 weeks.
Period: Overall Study
Arm/Group | Cohort 1 Tulisokibart | Cohort 1 Placebo | Cohort 2 Tulisokibart | Cohort 2 Placebo
Started | 68 | 67 | 22 | 21
Treated | 68 | 67 | 22 | 21
Completed | 0 | 0 | 0 | 0
Not Completed | 68 | 67 | 22 | 21
Not completed — Adverse Event | 0 | 2 | 0 | 1
Not completed — Lack of Efficacy | 0 | 2 | 0 | 0
Not completed — Prohibited Medication | 0 | 1 | 0 | 0
Not completed — Ongoing | 68 | 60 | 22 | 20
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Tulisokibart | Cohort 1 Placebo | Cohort 2 Tulisokibart | Cohort 2 Placebo | Total
Number analyzed (Participants) | 68 | 67 | 22 | 21 | 178
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.4 (14.4) | 42.2 (16.3) | 38.1 (18.2) | 38.5 (11.4) | 40.6 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 29 | 10 | 4 | 77
  Male | 34 | 38 | 12 | 17 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 1 | 1 | 8
  Not Hispanic or Latino | 60 | 62 | 19 | 19 | 160
  Unknown or Not Reported | 4 | 3 | 2 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 2
  White | 65 | 57 | 17 | 20 | 159
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 2 | 6 | 3 | 1 | 12
CDx+/CDx- [Number; unit: Participants] — CDx+ or CDx- status was determined by a genetic-based companion diagnostic (CDx) test governed by a protocol prespecified algorithm to identify participants who are predisposed for increased expression of Tumor necrosis factor-like cytokine 1A (TL1A) and therefore potentially more likely to respond to tulisokibart.
  Participants
    CDx+ | 16 | 16 | 22 | 21 | 75
    CDx- | 52 | 51 | 0 | 0 | 103
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Weight (kg) / [Height (m)]^2] — BMI was calculated for participants who had data from height and weight measurements collected at screening and Week 12/End of Treatment using the following formula: BMI = Weight (kg) / [Height (m)]^2. Population: BMI is reported for participants who had data available.
  Weight (kg) / [Height (m)]^2
    number analyzed (Participants) | 68 | 67 | 22 | 20 | 177
    (all) | 25.71 (7.029) | 25.52 (5.033) | 25.11 (4.539) | 26.37 (5.518) | 25.63 (5.845)
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Mean height of participants Population: Mean height is reported for participants who had data available.
  Centimeters (cm)
    number analyzed (Participants) | 68 | 67 | 22 | 20 | 177
    (all) | 169.91 (9.798) | 172.61 (9.185) | 172.31 (8.729) | 173.26 (8.418) | 171.61 (9.317)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Mean weight of participants
  Kilograms (kg) | 73.89 (19.653) | 76.59 (18.482) | 74.62 (14.985) | 79.36 (14.984) | 75.64 (18.135)
Duration of Ulcerative Colitis (UC) [Mean (Standard Deviation); unit: Years] — Mean duration of UC in years in participants
  Years | 6.680 (6.3766) | 6.277 (6.1942) | 5.911 (4.0708) | 10.351 (6.8957) | 6.866 (6.2239)
Time Since Symptom Onset [Mean (Standard Deviation); unit: Years] — Mean time in years for UC symptom onset in participants Population: Data for UC symptom onset duration was reported for participants who had data available.
  Years
    number analyzed (Participants) | 66 | 63 | 22 | 20 | 171
    (all) | 7.422 (6.2596) | 6.661 (5.7342) | 6.221 (4.0697) | 11.367 (6.5819) | 7.449 (6.0077)
Extent of UC [Count of Participants; unit: Participants] — Participant's extent of UC is classified as proctosigmoiditis, left sided colitis, or pancolitis.
  Participants
    Proctosigmoiditis | 2 | 7 | 2 | 1 | 12
    Left sided colitis | 35 | 28 | 10 | 8 | 81
    Pancolitis | 31 | 32 | 10 | 12 | 85
Current smoking status [Count of Participants; unit: Participants] — Participants smoking status is recorded as never, current, or former.
  Participants
    Never | 39 | 45 | 13 | 11 | 108
    Current | 9 | 3 | 3 | 0 | 15
    Former | 20 | 19 | 6 | 10 | 55
Baseline Endoscopic Score [Count of Participants; unit: Participants] — Baseline endoscopic score is part of the 3-component Modified Mayo Score (MMS), which is composed of endoscopic assessment, rectal bleeding, and stool frequency subscores with each of the components ranging from 0 to 3, with higher scores indicating more severe disease. The baseline endoscopy performed during screening is a malignancy surveillance colonoscopy for participants who have a diagnosis of UC for ≥ 7 years and have not had a screening colonoscopy for > 1 year.
  Participants
    Score of 2 | 22 | 14 | 3 | 9 | 48
    Score of 3 | 46 | 53 | 19 | 12 | 130
Baseline 3-Component Modified Mayo Score [Mean (Standard Deviation); unit: Score] — The 3-component MMS ranges from 0 to 9 and is composed of endoscopic assessment, rectal bleeding, and stool frequency subscores with each of the components ranging from 0 to 3, with higher scores indicating more severe disease. Population: The 3-component MMS is reported for all participants who had data available.
  Score
    number analyzed (Participants) | 68 | 67 | 21 | 21 | 177
    (all) | 6.9 (1.21) | 7.1 (1.10) | 7.1 (1.01) | 6.7 (1.27) | 7.0 (1.16)
Baseline Total Modified Mayo Score [Mean (Standard Deviation); unit: Score] — The Total MMS ranges from 0-12 and is composed of endoscopic assessment, rectal bleeding, stool frequency and physician global assessment (PGA) subscores with each of the components ranging from 0 to 3, with higher scores indicating more severe disease. Population: Total MMS is reported for all participants who had data available.
  Score
    number analyzed (Participants) | 68 | 67 | 21 | 21 | 177
    (all) | 9.1 (1.49) | 9.4 (1.29) | 9.3 (1.10) | 8.9 (1.59) | 9.2 (1.39)
Baseline High sensitivity C-reactive protein (hsCRP) [Mean (Standard Deviation); unit: mg/L] — hsCRP is an inflammatory biomarker and was obtained via blood and serum samples from participants. Population: Baseline hsCRP is reported for participants who had data available.
  mg/L
    number analyzed (Participants) | 67 | 67 | 22 | 21 | 177
    (all) | 10.162 (19.1910) | 10.022 (13.7709) | 10.754 (13.9272) | 10.155 (16.6271) | 10.182 (16.2430)
Concomitant UC Medication Use [Count of Participants; unit: Participants] — Concomitant medications are classified according to anatomical therapeutic chemical (ATC) drug classes using the World Health Organization (WHO) drug dictionary version March 2020 or newer. Medications are classified as oral corticosteroid, immunomodulator, or aminosalicylate. Prior medications are defined as the medication that started and stopped before the first dosing date. Only medications where the stop date is prior to the first dosing date were considered prior.
  Participants
    Oral Corticosteroid | 35 | 38 | 8 | 7 | 88
    Immunomodulator | 8 | 11 | 2 | 0 | 21
    Aminosalicylate | 44 | 45 | 16 | 14 | 119
Prior Treatment for UC [Count of Participants; unit: Participants] — Prior medications are classified according to ATC drug classes using the WHO drug dictionary version March 2020 or newer. Medications are classified as corticosteroid, immunomodulators, biologic or biologic-like.
  Participants
    Corticosteroid | 51 | 58 | 17 | 16 | 142
    Immunomodulators | 22 | 28 | 6 | 6 | 62
    Biologic/Biologic-Like Use (stratification) Yes | 35 | 35 | 12 | 12 | 94
    Biologic/Biologic-Like Use (stratification) No | 33 | 32 | 10 | 9 | 84
    Biologic/Biologic-Like Use (Prior Medications) Yes | 32 | 32 | 13 | 10 | 87
    Biologic/Biologic-Like Use (Prior Medications) No | 36 | 35 | 9 | 11 | 91

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Cohort 1 Achieving Clinical Remission
Description: The 3-component Modified Mayo Score (MMS) ranges from 0 to 9 and is composed of endoscopic assessment, rectal bleeding (RB), and stool frequency (SF) subscores with each of the components ranging from 0 to 3, with higher scores indicating more severe disease. Clinical remission is defined as endoscopic subscore of 0 or 1, RB subscore of 0, and SF subscore of 0 or 1 and not greater than baseline. Per protocol participants in Cohort 1 were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: All randomized participants in Cohort 1 who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 Tulisokibart | Cohort 1 Placebo
Number analyzed (Participants) | 68 | 67
Percentage of participants | 26.5 | 1.5
Statistical Analysis 1: Comparison: Cohort 1 Tulisokibart vs Cohort 1 Placebo; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; P-value is computed using Cochran-Mantel Haenszel (CMH) test with stratification factors of biologic status and CDx status; Risk Difference (RD) = 25.0, 95% CI 2-sided [11.8 to 36.5] — 95% CI is estimated using Newcombe method for risk difference

2. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. Reported adverse experiences used the Common Terminology for Adverse Events (CTCAE) Version 4.0. Per protocol, adverse events are reported by treatment with tulisokibart or placebo regardless of assigned cohort. Participants received identical treatment regiments regardless of cohort. The percentage of participants who experienced at least one AE is reported.
Time Frame: Up to ~14 weeks
Population: All randomized participants who received at least one dose of study intervention regardless of assigned cohort
Measure: Number; unit: Percentage of participants
Groups:
- All Cohorts (Cohort 1 & Cohort 2) Tulisokibartt: Participants received tulisokibart administered by intravenous (IV) infusion at 1000 mg on Day 1, Week 0 and 500 mg on the first day of Weeks 2, 6, and 10 regardless of cohort. After the completion of the 12-week induction, all participants have the option to continue in the open-label extension for up to 170 weeks.
- All Cohorts (Cohort 1 & Cohort 2) Placebo: Participants received placebo administered by intravenous (IV) infusion on Day 1, Week 0 and the first day of Weeks 2, 6, and 10 regardless of cohort. After the completion of the 12-week induction, all participants have the option to continue in the open-label extension for up to 170 weeks.
Arm/Group | All Cohorts (Cohort 1 & Cohort 2) Tulisokibartt | All Cohorts (Cohort 1 & Cohort 2) Placebo
Number analyzed (Participants) | 90 | 88
Percentage of participants | 45.6 | 43.2

3. Primary Outcome: Percentage of Participants Who Discontinued Due to an AE
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. Reported adverse experiences used the Common Terminology for Adverse Events (CTCAE) Version 4.0. Per protocol, adverse events are reported by treatment with tulisokibart or placebo regardless of assigned cohort. Participants received identical treatment regiments regardless of cohort. The percentage of participants who discontinued due to an AE is reported.
Time Frame: Up to ~14 weeks
Population: All randomized participants who received at least one dose of study intervention regardless of assigned cohort
Measure: Number; unit: Percentage of participants
Groups:
- All Cohorts (Cohort 1 & Cohort 2) Tulisokibart: Participants received tulisokibart administered by intravenous (IV) infusion at 1000 mg on Day 1, Week 0 and 500 mg on the first day of Weeks 2, 6, and 10 regardless of cohort. After the completion of the 12-week induction, all participants have the option to continue in the open-label extension for up to 170 weeks.
Arm/Group | All Cohorts (Cohort 1 & Cohort 2) Tulisokibart | All Cohorts (Cohort 1 & Cohort 2) Placebo
Number analyzed (Participants) | 90 | 88
Percentage of participants | 1.1 | 3.4

4. Secondary Outcome: Percentage of Participants in Cohort 1 With Endoscopic Improvement
Description: The 3-component MMS ranges from 0 to 9 and is composed of endoscopic assessment, RB, and SF subscores with each of the components ranging from 0 to 3, with higher scores indicating more severe disease. Endoscopic improvement is defined by endoscopy subscore of the MMS of ≤ 1 with no friability. Per protocol participants in Cohort 1 were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: All randomized participants in Cohort 1 who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 Tulisokibart | Cohort 1 Placebo
Number analyzed (Participants) | 68 | 67
Percentage of participants | 36.8 | 6.0
Statistical Analysis 1: Comparison: Cohort 1 Tulisokibart vs Cohort 1 Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 30.8, 95% CI 2-sided [17.4 to 43.2] — 95% CI is estimated using Newcombe method for risk difference

5. Secondary Outcome: Percentage of Participants in Cohort 1 Achieving Clinical Response
Description: The 3-component MMS ranges from 0 to 9 and is composed of endoscopic assessment, RB, and SF subscores with each of the components ranging from 0 to 3, with higher scores indicating more severe disease. Clinical response is defined as a reduction from Baseline ≥ 2 points and ≥ 30% in 3-component Modified Mayo Score, accompanied by a reduction ≥ 1 in RB subscore or absolute RB subscore ≤ 1. Per protocol participants in Cohort 1 were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: All randomized participants in Cohort 1 who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 Tulisokibart | Cohort 1 Placebo
Number analyzed (Participants) | 68 | 67
Percentage of participants | 66.2 | 22.4
Statistical Analysis 1: Comparison: Cohort 1 Tulisokibart vs Cohort 1 Placebo; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 43.8, 95% CI 2-sided [27.4 to 56.9] — 95% CI is estimated using Newcombe method for risk difference

6. Secondary Outcome: Percentage of Participants Who Were CDx+ (Cohorts 1 + 2) With Clinical Remission
Description: The 3-component MMS ranges from 0 to 9 and is composed of endoscopic assessment, RB, and SF subscores with each of the components ranging from 0 to 3, with higher scores indicating more severe disease. Clinical remission is defined as endoscopic subscore of 0 or 1, RB subscore of 0, and SF subscore of 0 or 1 and not greater than baseline. Per protocol participants who were CDx+ (Cohort 1 + Cohort 2) were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: All randomized participants who were CDx+ (Cohorts 1 + 2), who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Groups:
- CDx+ (Cohort 1 & Cohort 2) Tulisokibart: Participants who were CDx+ in Cohort 1 and Cohort 2 received tulisokibart administered by intravenous (IV) infusion at 1000 mg on Day 1, Week 0 and 500 mg on the first day of Weeks 2, 6, and 10. After the completion of the 12-week induction, all participants have the option to continue in the open-label extension for up to 170 weeks.
- CDx+ (Cohort 1 & Cohort 2) Placebo: Participants who were CDx+ in Cohort 1 and Cohort 2 received placebo administered by intravenous (IV) infusion on Day 1, Week 0 and the first day of Weeks 2, 6, and 10. After the completion of the 12-week induction, all participants have the option to continue in the open-label extension for up to 170 weeks.
Arm/Group | CDx+ (Cohort 1 & Cohort 2) Tulisokibart | CDx+ (Cohort 1 & Cohort 2) Placebo
Number analyzed (Participants) | 38 | 37
Percentage of participants | 31.6 | 10.8
Statistical Analysis 1: Comparison: CDx+ (Cohort 1 & Cohort 2) Tulisokibart vs CDx+ (Cohort 1 & Cohort 2) Placebo; Test type: Superiority; p = 0.0224, Cochran-Mantel-Haenszel; P-value is computed using Cochran-Mantel Haenszel (CMH) test with stratification factor of biologic status; Risk Difference (RD) = 20.8, 95% CI [2.1 to 37.9] — 95% CI is estimated using Newcombe method for risk difference

7. Secondary Outcome: Percentage of Participants in Cohort 1 With Symptomatic Remission
Description: RB, and SF subscores each range from 0 to 3, with higher scores indicating more severe disease. Symptomatic remission is defined as participants with SF subscore = 0 and RB subscore = 0. The percentage of participants who achieved symptomatic remission is presented. Per protocol participants in Cohort 1 were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: All randomized participants in Cohort 1 who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 Tulisokibart | Cohort 1 Placebo
Number analyzed (Participants) | 68 | 67
Percentage of participants | 19.1 | 6.0
Statistical Analysis 1: Comparison: Cohort 1 Tulisokibart vs Cohort 1 Placebo; Test type: Superiority; p = 0.0223, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 13.1, 95% CI [1.8 to 24.6] — 95% CI is estimated using Newcombe method for risk difference

8. Secondary Outcome: Percentage of Participants in Cohort 1 With Histologic Improvement
Description: Histologic improvement is defined as Geboes score ≤ 3.1. The Geboes histologic index includes 7 histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades from 0 to 5, with each grade of the score divided into 4 or 5 subcategories; the score ranges from 0.0 to 5.4. A higher score indicates more severe disease. Per protocol participants in Cohort 1 were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: All randomized participants in Cohort 1 who received at least one dose of study intervention and had baseline and Week 12 Geboes scores
Measure: Number; unit: Percentage
Arm/Group | Cohort 1 Tulisokibart | Cohort 1 Placebo
Number analyzed (Participants) | 65 | 57
Percentage | 46.2 | 17.5
Statistical Analysis 1: Comparison: Cohort 1 Tulisokibart vs Cohort 1 Placebo; Test type: Superiority; p = 0.0009, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 28.6, 95% CI [12.1 to 42.9] — 95% CI is estimated using Newcombe method for risk difference

9. Secondary Outcome: Percentage of Participants in Cohort 1 With Histologic-endoscopic Mucosal Improvement
Description: Histologic-endoscopic mucosal improvement is defined as a Geboes score ≤ 3.1 and endoscopy subscore of the MMS ≤ 1 with no friability. The Geboes histologic index includes 7 histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades from 0 to 5, with each grade of the score divided into 4 or 5 subcategories; the score ranges from 0.0 to 5.4. The endoscopic subscore of the MMS ranges from 0-3. For both scales a higher score indicates more severe disease. Per protocol participants in Cohort 1 were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 Tulisokibart | Cohort 1 Placebo
Number analyzed (Participants) | 65 | 57
Percentage of participants | 30.8 | 3.5
Statistical Analysis 1: Comparison: Cohort 1 Tulisokibart vs Cohort 1 Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 27.3, 95% CI [14.3 to 39.6] — 95% CI is estimated using Newcombe method for risk difference

10. Secondary Outcome: Percentage of Participants Who Were CDx+ (Cohorts 1 + 2) With Endoscopic Improvement
Description: The 3-component MMS ranges from 0 to 9 and is composed of endoscopic assessment, RB, and SF subscores with each of the components ranging from 0 to 3, with higher scores indicating more severe disease. Endoscopic improvement is defined by endoscopy subscore of MMS of ≤ 1 with no friability. Per protocol participants who were CDx+ (Cohort 1 + Cohort 2) were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: All randomized participants who were CDx+ (Cohorts 1 + 2), who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | CDx+ (Cohort 1 & Cohort 2) Tulisokibart | CDx+ (Cohort 1 & Cohort 2) Placebo
Number analyzed (Participants) | 38 | 37
Percentage of participants | 36.8 | 18.9
Statistical Analysis 1: Comparison: CDx+ (Cohort 1 & Cohort 2) Tulisokibart vs CDx+ (Cohort 1 & Cohort 2) Placebo; Test type: Superiority; Risk Difference (RD) = 17.9, 95% CI [-2.4 to 36.4] — 95% CI is estimated using Newcombe method for risk difference

11. Secondary Outcome: Percentage of Participants Who Were CDx+ (Cohorts 1 + 2) With Clinical Response
Description: The 3-component MMS ranges from 0 to 9 and is composed of endoscopic assessment, RB, and SF subscores with each of the components ranging from 0 to 3, with higher scores indicating more severe disease. Clinical response is defined by reduction from Baseline ≥ 2 points and ≥ 30% in 3-component Modified Mayo Score, accompanied by a reduction ≥ 1 in RB subscore or absolute RB subscore ≤ 1. Per protocol participants who were CDx+ (Cohort 1 + Cohort 2) were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: All randomized participants who were CDx+ (Cohorts 1 + 2), who received at least one dose of study intervention
Measure: Number; unit: Percentage of Participants
Arm/Group | CDx+ (Cohort 1 & Cohort 2) Tulisokibart | CDx+ (Cohort 1 & Cohort 2) Placebo
Number analyzed (Participants) | 38 | 37
Percentage of Participants | 55.3 | 32.4
Statistical Analysis 1: Comparison: CDx+ (Cohort 1 & Cohort 2) Tulisokibart vs CDx+ (Cohort 1 & Cohort 2) Placebo; Test type: Superiority; Risk Difference (RD) = 22.8, 95% CI [0.4 to 42.2] — 95% CI is estimated using Newcombe method for risk difference

12. Secondary Outcome: Percentage of Participants Who Were CDx+ (Cohorts 1 + 2) With Symptomatic Remission
Description: RB, and SF subscores each range from 0 to 3, with higher scores indicating more severe disease. Symptomatic remission is defined as participants with SF subscore = 0 and RB subscore = 0. The percentage of participants who achieved symptomatic remission is presented. Per protocol participants who were CDx+ (Cohort 1 + Cohort 2) were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: All randomized participants who were CDx+ (Cohorts 1 + 2), who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | CDx+ (Cohort 1 & Cohort 2) Tulisokibart | CDx+ (Cohort 1 & Cohort 2) Placebo
Number analyzed (Participants) | 38 | 37
Percentage of participants | 21.1 | 10.8
Statistical Analysis 1: Comparison: CDx+ (Cohort 1 & Cohort 2) Tulisokibart vs CDx+ (Cohort 1 & Cohort 2) Placebo; Test type: Superiority; Risk Difference (RD) = 10.2, 95% CI [-6.9 to 26.9] — 95% CI is estimated using Newcombe method for risk difference

13. Secondary Outcome: Percentage of Participants Who Were CDx+ (Cohorts 1 + 2) With Histologic Improvement
Description: Histologic improvement is defined as Geboes score ≤ 3.1. The Geboes histologic index includes 7 histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades from 0 to 5, with each grade of the score divided into 4 or 5 subcategories; the score ranges from 0.0 to 5.4. A higher score indicates more severe disease. Per protocol participants who were CDx+ (Cohorts 1 + 2) were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: All randomized participants who were CDx+ (Cohorts 1 + 2), who received at least one dose of study intervention and had baseline and Week 12 data for Geboes Scores
Measure: Number; unit: Percentage of participants
Arm/Group | CDx+ (Cohort 1 & Cohort 2) Tulisokibart | CDx+ (Cohort 1 & Cohort 2) Placebo
Number analyzed (Participants) | 36 | 30
Percentage of participants | 55.6 | 26.7
Statistical Analysis 1: Comparison: CDx+ (Cohort 1 & Cohort 2) Tulisokibart vs CDx+ (Cohort 1 & Cohort 2) Placebo; Test type: Superiority; Risk Difference (RD) = 28.9, 95% CI [5.0 to 48.3] — 95% CI is estimated using Newcombe method for risk difference

14. Secondary Outcome: Percentage of Participants Who Were CDx+ (Cohorts 1 + 2) With Histologic-endoscopic Mucosal Improvement
Description: Histologic-endoscopic mucosal improvement is defined as a Geboes score ≤ 3.1 and endoscopy subscore of the MMS ≤ 1 with no friability. The Geboes histologic index includes 7 histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades from 0 to 5, with each grade of the score divided into 4 or 5 subcategories; the score ranges from 0.0 to 5.4. The endoscopic subscore of the MMS ranges from 0-3. For both scales a higher score indicates more severe disease. Per protocol participants who were CDx+ (Cohorts 1 + 2) were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: All participants who were CDx+ (Cohorts 1 + 2), who received at least one dose of study intervention and had baseline and Week 12 data for Geboes Scores
Measure: Number; unit: Percentage of participants
Arm/Group | CDx+ (Cohort 1 & Cohort 2) Tulisokibart | CDx+ (Cohort 1 & Cohort 2) Placebo
Number analyzed (Participants) | 36 | 30
Percentage of participants | 38.9 | 16.7
Statistical Analysis 1: Comparison: CDx+ (Cohort 1 & Cohort 2) Tulisokibart vs CDx+ (Cohort 1 & Cohort 2) Placebo; Test type: Superiority; Risk Difference (RD) = 22.2, 95% CI 2-sided [0.2 to 41.0] — 95% CI is estimated using Newcombe method for risk difference

15. Secondary Outcome: Percentage of Participants in Cohort 1 With Histologic-endoscopic Mucosal Healing
Description: Histologic-endoscopic mucosal improvement is defined as Geboes score ≤ 2B.1 and endoscopy subscore of MMS ≤ 1 with no friability. The Geboes histologic index includes 7 histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades from 0 to 5, with each grade of the score divided into 4 or 5 subcategories; the score ranges from 0.0 to 5.4. The endoscopic subscore of the MMS ranges from 0-3. For both scales a higher score indicates more severe disease. Per protocol participants in Cohort 1 were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: All randomized participants in Cohort 1 who received at least one dose of study intervention and had baseline and Week 12 data for Geboes Scores
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 Tulisokibart | Cohort 1 Placebo
Number analyzed (Participants) | 65 | 57
Percentage of participants | 30.8 | 3.5
Statistical Analysis 1: Comparison: Cohort 1 Tulisokibart vs Cohort 1 Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 27.3, 95% CI 2-sided [14.3 to 39.6] — 95% CI is estimated using Newcombe method for risk difference

16. Secondary Outcome: Percentage of Participants Who Were CDx+ (Cohorts 1 + 2) With Histologic-endoscopic Mucosal Healing
Description: Histologic-endoscopic mucosal improvement is defined as Geboes score ≤ 2B.1 and endoscopy subscore of MMS ≤ 1 with no friability. The Geboes histologic index includes 7 histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades from 0 to 5, with each grade of the score divided into 4 or 5 subcategories; the score ranges from 0.0 to 5.4. The endoscopic subscore of the MMS ranges from 0-3. For both scales a higher score indicates more severe disease. Per protocol participants who were CDx+ (Cohorts 1 + 2) were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | CDx+ (Cohort 1 & Cohort 2) Tulisokibart | CDx+ (Cohort 1 & Cohort 2) Placebo
Number analyzed (Participants) | 36 | 30
Percentage of participants | 38.9 | 16.7
Statistical Analysis 1: Comparison: CDx+ (Cohort 1 & Cohort 2) Tulisokibart vs CDx+ (Cohort 1 & Cohort 2) Placebo; Test type: Superiority; Risk Difference (RD) = 22.2, 95% CI [0.2 to 41.0] — 95% CI is estimated using Newcombe method for risk difference

17. Secondary Outcome: Percentage of Participants in Cohort 1 With an Inflammatory Bowel Disease Questionnaire (IBDQ) Response
Description: IBDQ is a self-administered, disease-specific Health-Related Quality of Life (HRQOL) instrument for subjects with IBD. The IBDQ covers 4 dimensions and 32 questions: bowel symptoms, systemic symptoms, emotional function, and social function. Items are scored on a 7-point Likert scale (1 = all of the time and 7 = none of the time), for a total global score in the range 32 to 224 (with higher scores indicating better HRQOL). IBDQ response, as defined by ≥ 16-point increase from Baseline at Week 12. Per protocol participants in Cohort 1 were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: All randomized participants in Cohort 1 who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 Tulisokibart | Cohort 1 Placebo
Number analyzed (Participants) | 68 | 67
Percentage of participants | 82.4 | 49.3
Statistical Analysis 1: Comparison: Cohort 1 Tulisokibart vs Cohort 1 Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 33.1, 95% CI [17.2 to 46.8] — 95% CI is estimated using Newcombe method for risk difference

18. Secondary Outcome: Percentage of Participants Who Are CDx+ (Cohorts 1 + 2) Who Had an IBDQ Response
Description: IBDQ is a self-administered, disease-specific Health-Related Quality of Life (HRQOL) instrument for subjects with IBD. The IBDQ covers 4 dimensions and 32 questions: bowel symptoms, systemic symptoms, emotional function, and social function. Items are scored on a 7-point Likert scale (1 = all of the time and 7 = none of the time), for a total global score in the range 32 to 224 (with higher scores indicating better HRQOL). IBDQ response, as defined by ≥ 16-point increase from Baseline at Week 12. Per protocol participants who were CDx+ (Cohorts 1 + 2) were analyzed for this outcome measure.
Time Frame: Baseline and Week 12
Population: All randomized participants who were CDx+ (Cohorts 1 + 2), who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | CDx+ (Cohort 1 & Cohort 2) Tulisokibart | CDx+ (Cohort 1 & Cohort 2) Placebo
Number analyzed (Participants) | 38 | 37
Percentage of participants | 76.3 | 56.8
Statistical Analysis 1: Comparison: CDx+ (Cohort 1 & Cohort 2) Tulisokibart vs CDx+ (Cohort 1 & Cohort 2) Placebo; Test type: Superiority; Risk Difference (RD) = 19.6, 95% CI [-1.7 to 38.7] — 95% CI is estimated using Newcombe method for risk difference

19. Primary Outcome: Percentage of Participants Who Had One or More Serious Adverse Events
Description: Reported adverse experiences used the Common Terminology for Adverse Events (CTCAE) Version 4.0. Serious adverse events are defined as: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living (ADL), Life-threatening consequences; urgent intervention indicated, and death. Per protocol, adverse events are reported by treatment with tulisokibart or placebo regardless of assigned cohort. Participants received identical treatment regiments regardless of cohort. The percentage of participants experiencing a serious AE are presented.
Time Frame: Up to ~14 weeks
Population: All randomized participants who received at least one dose of study intervention regardless of assigned cohort
Measure: Number; unit: Percentage of participants
Arm/Group | All Cohorts (Cohort 1 & Cohort 2) Tulisokibart | All Cohorts (Cohort 1 & Cohort 2) Placebo
Number analyzed (Participants) | 90 | 88
Percentage of participants | 1.1 | 8.0

ADVERSE EVENTS:
Time Frame: Death and Adverse Events up to ~14 weeks.
Description: Per protocol death and adverse events are grouped by treatment or placebo irrespective of cohort. Participants in Cohorts 1 and 2 received identical treatment.
Arm/Group | All Cohorts (Cohort 1 & Cohort 2) Tulisokibart | All Cohorts (Cohort 1 & Cohort 2) Placebo
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/88
Serious Adverse Events (participants affected / at risk) | 1/90 | 7/88
Other Adverse Events (participants affected / at risk) | 5/90 | 4/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Cohorts (Cohort 1 & Cohort 2) Tulisokibart (N=90) | All Cohorts (Cohort 1 & Cohort 2) Placebo (N=88)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 5 (5)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Cohorts (Cohort 1 & Cohort 2) Tulisokibart (N=90) | All Cohorts (Cohort 1 & Cohort 2) Placebo (N=88)
COVID-19 (Infections and infestations) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information concerning the product subsequently generated from this study (such as patent applications, formulae, manufacturing processes, basic scientific data, or formulation information supplied to the Investigator by the Sponsor and not previously published) is considered confidential by and shall remain the sole property of the Sponsor. The Investigator agrees not to use it for other purposes without the Sponsor's written consent.

DOCUMENTS (2):
  • Study Protocol (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT04996797/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT04996797/SAP_001.pdf